CLINICAL TRIAL: NCT04962152
Title: To Explore the Effects of Naldebain Combined With Thoracic Paravertebral Block in Video-assisted Thoracoscopic Surgery.
Brief Title: Naldebain and Video-assisted Thoracoscopic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20210087
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-07

CONDITIONS: Analgesia; Nausea and Vomiting, Postoperative; Itching; Injection Site Reaction; Satisfaction, Patient
MeSH Terms: conditions — Agnosia; Postoperative Nausea and Vomiting; Pruritus; Injection Site Reaction; Patient Satisfaction | interventions — Sesame Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Naldebain (Experimental): ultrasound-guided intramuscular injection of Naldebain 150mg after the induction anesthesia immediately
  Interventions: Drug: Nalbuphine Sebacate or Sesame oil (placebo)
- Group Placebo (Placebo Comparator): ultrasound-guided intramuscular injection of sesame oil (placebo) 2mL after the induction anesthesia immediately
  Interventions: Drug: Nalbuphine Sebacate or Sesame oil (placebo)

INTERVENTIONS:
Drug: Nalbuphine Sebacate or Sesame oil (placebo) — ultrasound-guided intramuscular injection after the induction of anesthesia immediately
  Other Names: Naldebain ER

SUMMARY:
To evaluate the postoperative analgesic effect of combined use of Naldebain® and thoracic paravertebral block in thoracoscopic surgery

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) can be associated with stronger postoperative pain than is commonly believed. Pain control after thoracic surgery is important because increased acute pain has been shown to increase the incidence of chronic pain, and untreated pain may lead to increased morbidity. It is generally accepted to introduce multimodal analgesic strategies based on regional blockade, opioids and non-steroidal anti-inflammatory drugs.

Paravertebral block (PVB) involves the injection of local anesthetic into a wedge-shaped space lateral to the spinal nerves as they emerge from intervertebral foramina. It produces ipsilateral somatosensory and sympathetic nerve blockade effective for anesthesia as well as for management of pain of unilateral origin from the chest and abdomen. So far, thoracic paravertebral block (TPVB) is the most common technique used for patients undergoing VATS. TPVB may be useful after VATS because a single injection of local anesthesia may provide effective analgesia for the intense short-duration pain that patients experience.

Nalbuphine sebacate (Naldebain®) is a long-acting prodrug of nalbuphine developed for meeting the unmet medical need of long-acting analgesics. It is a synthetic opioid agonist-antagonist analgesic of the phenanthrene series. It is chemically related to both the widely used opioid antagonist, naloxone, and the potent opioid analgesic, oxymorphone. The currently proposed clinical use of nalbuphine sebacate is a single dose of Naldebain® administered intramuscularly approximately 24 h prior to the planned surgery for pain relief.

The purpose of this study is to determine the safety and efficacy of TPVB combined with a single dose of intramuscular Naldebain® administered preoperatively to patients scheduled to undergo VATS.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subject's age: 20~65 years old
* 2) American Society of Anesthesiologists (ASA) Physical Status classification: I~III
* 3) Patients who need postoperative pain relief due to thoracoscopic surgery

Exclusion Criteria:

* 1. The patient suffers from a communication disorder
* 2. The patient has coagulopathy
* 3. Sick with obvious heart, lung, liver or kidney disease
* 4. The patient's body mass index is less than 18.5 or greater than 35
* 5. Pregnant patients
* 6. Patients who took opioids for more than three weeks before surgery
* 7. Patients with contraindications to local anesthesia
* 8. Patients with a history of chronic pain
* 9. Patients with a history of drug allergy to Naldebain

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-05-07 (Estimated); Study Completion 2024-05-07 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesic effect | During the first one hour in the recovery room, the pain intensity was evaluated every 15 minutes.
  Use the visual analogue scale (VAS) score to assess the degree of pain after surgery
postoperative analgesic effect | the pain intensity was evaluated at 3 hours after surgery.
  Use the visual analogue scale (VAS) score to assess the degree of pain after surgery
postoperative analgesic effect | the pain intensity was evaluated at 6 hours after surgery.
  Use the visual analogue scale (VAS) score to assess the degree of pain after surgery
postoperative analgesic effect | the pain intensity was evaluated at 12 hours after surgery.
  Use the visual analogue scale (VAS) score to assess the degree of pain after surgery
postoperative analgesic effect | the pain intensity was evaluated at 24 hours after surgery.
  Use the visual analogue scale (VAS) score to assess the degree of pain after surgery
postoperative analgesic effect | the pain intensity was evaluated at 36 hours after surgery.
  Use the visual analogue scale (VAS) score to assess the degree of pain after surgery
postoperative analgesic effect | the pain intensity was evaluated at 48 hours after surgery.
  Use the visual analogue scale (VAS) score to assess the degree of pain after surgery
postoperative analgesic effect | the pain intensity was evaluated at 72 hours after surgery.
  Use the visual analogue scale (VAS) score to assess the degree of pain after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Te Hsu, MD, PhD, Principal Investigator — Department of anesthesiology, Kaohsiung Medical University Hospital
Locations (1):
- Department of Anesthesiology, Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Hsu HT, Ma CW, Chang PC, Kuo YW, Gau TP, Liu YW, Liu YC, Chou SH, Cheng KI. Effect of Dinalbuphine sebacate on postoperative multimodal analgesic strategy in video-assisted thoracoscopic surgery: a double-blind randomized controlled trial. BMC Anesthesiol. 2025 May 17;25(1):252. doi: 10.1186/s12871-025-03118-7. PMID 40382572